CLINICAL TRIAL: NCT05696015
Title: Impact of Telehealth Education After Hospital Discharge on the Self-care of Patients With Diabetes
Brief Title: Impact of Telehealth Education in Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Simone Brandi, Principal investigator, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 61722122.8.0000.0071
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: self care
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The randomized clinical trial.
Masking Description: Patients will be randomized using the Randomizer software into a group that will receive the telemonitoring intervention and a control group (which will only receive the hospital's standard hospital discharge instructions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard education (Active Comparator): Standard education group will be carried out at discharge, discharge orientation of the patient with diabetes and application of the Diabetes Self-Care Activity Questionnaire (QAD). For this group, a new contact will be made within 30 days after discharge, where the QAD will be applied again.
  Interventions: Behavioral: Standard education
- Amplied education (Experimental): Amplied education group will be performed at the time of discharge, guidance for discharge of patients with diabetes. This group will receive 3 contacts, the first will be carried out within 72 hours after discharge, the second contact within 10 days after the first contact and the third within 30 days after discharge, where diabetes education guidelines will be given to the patient in all contacts. At the time of discharge, and in the third contact, 30 days, the QAD will also be applied.
  Interventions: Behavioral: Ampiled Education

INTERVENTIONS:
Behavioral: Standard education — Without telehealth education, this group has only postdischarge education.
  Arms: Standard education
Behavioral: Ampiled Education — With telehealth education, in addition of discharge education.
  Arms: Amplied education

SUMMARY:
The goal of this clinical trial is to to evaluate the effectiveness of continuity of in-hospital care with the application of a structured telemonitoring protocol in self-care activities in patients with type 1 or type 2 Diabetes Mellitus or those who have an HbA1C level greater than or equal to 6.5% during hospitalization, regardless of the reason for hospitalization. The main question[s] it aims to answer are:

• Is telehealth education effective for improving self-care for type 1 or type 2 Diabetes Mellitus or those with an HbA1C level greater than or equal to 6.5% during hospitalization will be included, regardless of the reason for hospitalization? Participants will answer the Diabetes Self-Care Activity Questionnaire Researchers will compare patients in the intervention group, in addition to the hospital's standard hospital guidance, will receive an educational approach through structured telemonitoring, reinforcing and validating the points addressed in the face-to-face guidance, which are considered the foundations of self-care.

DETAILED DESCRIPTION:
This study have two groups of patients. Group 1 will be carried out at discharge, discharge orientation of the patient with diabetes and application of the Diabetes Self-Care Activity Questionnaire (QAD). For this group, a new contact will be made within 30 days after discharge, where the QAD will be applied again.

Group 2 will be performed at the time of discharge, guidance for discharge of patients with diabetes. This group will receive 3 contacts, the first will be carried out within 72 hours after discharge, the second contact within 10 days after the first contact and the third within 30 days after discharge, where diabetes education guidelines will be given to the patient in all contacts. At the time of discharge, and in the third contact, 30 days, the QAD will also be applied.

ELIGIBILITY:
Inclusion Criteria:

* patients who were hospitalized at Hospital Israelita Albert Einstein and included in the subcutaneous insulin protocol to control hyperglycemia
* patients monitored by the Diabetes Program, an institutional program that manages glycemic changes that occur within the institution.
* patients with type 1 or type 2 Diabetes Mellitus or those with an HbA1C level greater than or equal to 6.5% during hospitalization.

Exclusion Criteria:

* Patients not submitted to the first face-to-face educational approach required by protocol
* Patients discharged on the weekend or holidays

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-02 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline discharge orientation of the patient with diabetes and application of the Diabetes Self-Care Activity Questionnaire (QAD) at 30 days follow-up. (Standard education) | immediately pre and within 4 weeks post intervention
  The QAD instrument has six dimensions and 15 items for evaluating self-care with diabetes: "general diet" (two items), "specific diet" (three items), "physical activity" (two items) , "blood glucose monitoring" (two items), "foot care" (three items) and "medication use" (three items, used according to the medication regimen), in addition to three other items for the assessment of smoking . Patients answer how often (answers from 0 to 7) they performed the activities or behaviors in the seven days prior to completing the form.
  For the calculation of scores, the items of the specific food dimension that ask about the consumption of foods high in fat and sweets, the values must be inverted (7=0, 6=1, 5=2, 4=3, 3=4 , 2=5, 1=6 and 0=7). Scores are calculated by averaging the items that make up each dimension, with zero being the least desirable situation and seven being the most favorable.
Change from baseline discharge telehealth orientation and application of the Diabetes Self-Care Activity Questionnaire (QAD) at within 72 hours after discharge, 10 days after and within 30 days after discharge | immediately pre and within 72 hours after discharge, the second contact within 10 days after the first contact and the third within 30 days after discharge
  Patients in the intervention group, in addition to the hospital's standard hospital guidance, will receive an educational approach through structured telemonitoring, reinforcing and validating the points addressed in the face-to-face guidance, which are considered the foundations of self-care. Contacts will be made via video call by trained health professionals, who will provide care based on a script structured by the authors, assessing adherence to self-care. The American Association of Diabetes Educators ( 7 Self-Care Behaviors ™) ) is a structured evidence-based tool that allows, in addition to self-care assessment, educational intervention in the seven topics covered, which include: 1) healthy eating, 2) physical activity, 3) glycemic monitoring , 4) medication use, 5) problem solving, 6) healthy coping, and 7) risk reduction.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chrvala CA, Sherr D, Lipman RD. Diabetes self-management education for adults with type 2 diabetes mellitus: A systematic review of the effect on glycemic control. Patient Educ Couns. 2016 Jun;99(6):926-43. doi: 10.1016/j.pec.2015.11.003. Epub 2015 Nov 22. PMID 26658704
- [Result] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Result] Dong Y, Wang P, Dai Z, Liu K, Jin Y, Li A, Wang S, Zheng J. Increased self-care activities and glycemic control rate in relation to health education via Wechat among diabetes patients: A randomized clinical trial. Medicine (Baltimore). 2018 Dec;97(50):e13632. doi: 10.1097/MD.0000000000013632. PMID 30558051
- [Result] Ansari RM, Harris MF, Hosseinzadeh H, Zwar N. The Summary of an Urdu Version of Diabetes Self-Care Activities Measure: Psychometric Evaluation and Validation. J Prim Care Community Health. 2020 Jan-Dec;11:2150132720935292. doi: 10.1177/2150132720935292. PMID 32538255
- [Result] Frosch DL, Uy V, Ochoa S, Mangione CM. Evaluation of a behavior support intervention for patients with poorly controlled diabetes. Arch Intern Med. 2011 Dec 12;171(22):2011-7. doi: 10.1001/archinternmed.2011.497. Epub 2011 Oct 10. PMID 21986347
- [Result] Weinger K, Beverly EA, Smaldone A. Diabetes self-care and the older adult. West J Nurs Res. 2014 Oct;36(9):1272-98. doi: 10.1177/0193945914521696. Epub 2014 Feb 7. PMID 24510969
- [Result] Whitehouse CR, Long JA, Maloney LM, Daniels K, Horowitz DA, Bowles KH. Feasibility of Diabetes Self-Management Telehealth Education for Older Adults During Transitions in Care. Res Gerontol Nurs. 2020 May 1;13(3):138-145. doi: 10.3928/19404921-20191210-03. Epub 2019 Dec 13. PMID 31834415
- [Result] Ose D, Kamradt M, Kiel M, Freund T, Besier W, Mayer M, Krisam J, Wensing M, Salize HJ, Szecsenyi J. Care management intervention to strengthen self-care of multimorbid patients with type 2 diabetes in a German primary care network: A randomized controlled trial. PLoS One. 2019 Jun 12;14(6):e0214056. doi: 10.1371/journal.pone.0214056. eCollection 2019. PMID 31188825
- [Result] So CF, Chung JW. Telehealth for diabetes self-management in primary healthcare: A systematic review and meta-analysis. J Telemed Telecare. 2018 Jun;24(5):356-364. doi: 10.1177/1357633X17700552. Epub 2017 May 2. PMID 28463033